CLINICAL TRIAL: NCT00205036
Title: Impact of Calcium Supplements on Lumbar Spine Bone Mineral Density
Brief Title: Calcium DXA: Impact of Calcium Supplements on Lumbar Spine Bone Mineral Density
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: M-2004-1308
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Healthy

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
We, the investigators at the University of Wisconsin, hypothesized that ingesting calcium tablets prior to a spine bone density scan will not affect the bone mineral density as measured by dual energy x-ray absorptiometry (DXA).

DETAILED DESCRIPTION:
We hypothesized that ingesting calcium tablets prior to a spine bone density scan will not affect the bone mineral density as measured by DXA. To test this, 36 subjects ingested various calcium supplements after a spine DXA scan and were then scanned again 15, 30 and 45 minutes after ingestion. Subsequently a subset of 15 subjects had three spine scans performed for instrument precision and subsequently ingested a calcium tablet with scans 15 and 30 minute intervals after ingestion.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 years or older

Exclusion Criteria:

* Internal spinal hardware

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2005-01; Primary Completion 2005-10 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil C Binkley, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States